CLINICAL TRIAL: NCT02186093
Title: Clinical, Physiological and Prognostic Implication of Index of Microcirculatory Resistance
Brief Title: Clinical, Physiological and Prognostic Implication of Microvascular Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ulsan University Hospital (Other); Keimyung University (Other); Inje University (Other); Stanford University (Other); University of Glasgow (Other); Hospital San Carlos, Madrid (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1404-057-573
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2009-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Angina, Stable; Fractional Flow Reserve, Myocardial; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Korea: patients in South of Korea
- United Kingdom: patients in England
- Spain: patients in Spain
- United State of America: patients in USA

SUMMARY:
There are several physiologic parameters in evaluating cardiovascular disease. This study will reveal which parameter is the most proper value in predicting disease severity and risk factors of patients.

DETAILED DESCRIPTION:
Fractional Flow Reserve (FFR), index of microcirculatory resistance (IMR), and coronary flow reserve (CFR) will be measured in stable angina patients before coronary intervention.

Relationship between angiographic characteristics of patients and FFR, IMR, CFR will be analyzed. Comparison of risk factors and prognosis between parameters will be also analyzed. This study will evaluate that which parameter is correlate with disease severity and risk factors of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with stable angina
* FFR, IMR, CFR were measured before coronary intervention

Exclusion Criteria:

* Patients who have severe side effects or contraindication to hyperemic agents (ex. adenosine)
* Patients with hemodynamic instability
* elevation of cardiac enzymes, evidence of acute MI, or a culprit vessel of acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina
Sampling Method: Non-Probability Sample
Enrollment: 1197 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Spearman correlation coefficient between FFR, IMR, CFR and angiographic severity | during coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul national university hosptial; Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - Keimyung University Dongsan medical center, Daegu
  - Inje University Ilsan Paik Hospital, Goyang
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan

IPD SHARING:
Plan to Share IPD: No
Data will be available when requested after discussion in steering committee

REFERENCES:
- [Derived] Chung JH, Lee KE, Lee JM, Her AY, Kim CH, Choi KH, Song YB, Hahn JY, Kim HY, Choi JH, Garg S, Doh JH, Nam CW, Koo BK, Shin ES. Effect of Sex Difference of Coronary Microvascular Dysfunction on Long-Term Outcomes in Deferred Lesions. JACC Cardiovasc Interv. 2020 Jul 27;13(14):1669-1679. doi: 10.1016/j.jcin.2020.04.002. Epub 2020 Jun 24. PMID 32593698
- [Derived] Hoshino M, Hamaya R, Kanaji Y, Kanno Y, Hada M, Yamaguchi M, Sumino Y, Hirano H, Horie T, Usui E, Sugiyama T, Murai T, Lee T, Yonetsu T, Lee JM, Choi KH, Hwang D, Park J, Jung JH, Kim HY, Jung HW, Cho YK, Yoon HJ, Song YB, Hahn JY, Doh JH, Nam CW, Shin ES, Hur SH, Mejia-Renteria H, Lauri F, Goto S, Macaya F, McInerney A, Gravina G, Vera R, Gonzalo N, Jimenez-Quevedo P, Nunez-Gil I, Salinas P, Nombela-Franco L, Del Trigo M, Fernandez-Ortiz A, Macaya C, Koo BK, Escaned J, Kakuta T. Sex Differences in Long-Term Outcomes in Patients With Deferred Revascularization Following Fractional Flow Reserve Assessment: International Collaboration Registry of Comprehensive Physiologic Evaluation. J Am Heart Assoc. 2020 Feb 18;9(4):e014458. doi: 10.1161/JAHA.119.014458. Epub 2020 Feb 17. PMID 32063120
- [Derived] Lee SH, Choi KH, Lee JM, Hwang D, Rhee TM, Park J, Kim HK, Cho YK, Yoon HJ, Park J, Song YB, Hahn JY, Doh JH, Nam CW, Shin ES, Hur SH, Koo BK. Physiologic Characteristics and Clinical Outcomes of Patients With Discordance Between FFR and iFR. JACC Cardiovasc Interv. 2019 Oct 28;12(20):2018-2031. doi: 10.1016/j.jcin.2019.06.044. Epub 2019 Sep 25. PMID 31563683
- [Derived] Lee JM, Choi KH, Hwang D, Park J, Jung JH, Kim HY, Jung HW, Cho YK, Yoon HJ, Song YB, Hahn JY, Doh JH, Nam CW, Shin ES, Hur SH, Koo BK. Prognostic Implication of Thermodilution Coronary Flow Reserve in Patients Undergoing Fractional Flow Reserve Measurement. JACC Cardiovasc Interv. 2018 Aug 13;11(15):1423-1433. doi: 10.1016/j.jcin.2018.05.005. PMID 30093048
- [Derived] Lee JM, Jung JH, Hwang D, Park J, Fan Y, Na SH, Doh JH, Nam CW, Shin ES, Koo BK. Coronary Flow Reserve and Microcirculatory Resistance in Patients With Intermediate Coronary Stenosis. J Am Coll Cardiol. 2016 Mar 15;67(10):1158-1169. doi: 10.1016/j.jacc.2015.12.053. PMID 26965536
- [Derived] Lee JM, Layland J, Jung JH, Lee HJ, Echavarria-Pinto M, Watkins S, Yong AS, Doh JH, Nam CW, Shin ES, Koo BK, Ng MK, Escaned J, Fearon WF, Oldroyd KG. Integrated physiologic assessment of ischemic heart disease in real-world practice using index of microcirculatory resistance and fractional flow reserve: insights from the International Index of Microcirculatory Resistance Registry. Circ Cardiovasc Interv. 2015 Nov;8(11):e002857. doi: 10.1161/CIRCINTERVENTIONS.115.002857. PMID 26499500